CLINICAL TRIAL: NCT06020105
Title: Design and Development of a Nurse-led Program for the Management of Bariatric Surgery Patients - The NURLIFE Program
Brief Title: The NURLIFE Program for the Management of Bariatric Surgery Patients
Acronym: NURLIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Cláudia Mendes, Principal Investigator, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1635/22
Record Dates: First submitted 2023-08-25; First posted 2023-08-31 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Bariatric Surgery Candidate; Nurse-Patient Relations
Keywords: Case manager; e-health; Nurse case management; Bariatric surgery; Perioperative care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention will be a combination of consultations and face-to-face follow-ups, with teleconsultations, based on other observational and experimental studies. The intervention program includes monitoring for one year of patients enrolled in the bariatric surgery consultation, with criteria for surgeries.
  Interventions: Behavioral: NURLIFE
- Control Group (No Intervention): The control group will only carry out the assessments and will be offered the same intervention as the intervention group at the end of the intervention.

INTERVENTIONS:
Behavioral: NURLIFE — After the first consultation with the surgeon, the patients will be referred to the case manager, who will carry out the first face-to-face consultation, with consequent monitoring and clarification of identified needs, following the flowchart in figure 3, being referred to the different specialties, psychology, nutrition and nursing, fostering the case manager as the central pillar of the process, which will monitor each process individually, namely the number of consultations and necessary referrals.
  Arms: Intervention Group

SUMMARY:
to analyze the influence of the new intervention in the perioperative period and impact on several clinical and humanistic endpoints. In the evaluation phase, an experimental, controlled, and randomized study (RCT) will be developed, with an intervention group (IG) and a control group (CG). The CG will receive the usual care and the IG, will receive the intervention for an expected period of one year. This project aims to be the first study to investigate the effect of a long-term specialized case-management intervention (face-to-face and e-health) in patients who are candidates for bariatric surgery during all the perioperative periods

DETAILED DESCRIPTION:
The "nurse-led case-management" intervention program will allow to improve the management of the bariatric surgery process by patients in collaboration with the health team, with a view to improving health and adopting healthy lifestyles, which enhance better results. This intervention program is expected to be a mixed program with e-health technologies. Behavioural changes will be predictably one of the main objectives, with perception of the barriers and facilitators of them, from the perspective of training the patient for the physiological changes that result from the entire process of bariatric surgery. Thus, it is expected that the primary focus of the program will be health education and motivation for lifestyle changes, the promotion of healthy lifestyles and promotion of physical activity, with a view to improving anthropometric data and metabolic risk factors, as well as smoking cessation and alcoholic habits. As such, the contribution of a multidisciplinary team that is managed by a case-manager appears to be the most efficient intervention, and this activity aims to determine the set of procedures and their temporal sequence, the skills of the team, the flow of patients through the different elements of the team and the duration of the program.

ELIGIBILITY:
Inclusion Criteria:

* As inclusion criteria, patients should be enrolled for bariatric surgery at the hospital
* Agree to participate in the study

Exclusion Criteria:

* Surgical complications
* Psychiatric diseases and neurological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-01-02 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Body weight | 1 year
  scale
Height | 1 year
  stadiometer
cholesterol in mg/dl | 1 year
  Blood sample
Glucose in mg/dl | 1 year
  Blood sample
Mean blood pressure | 1 year
  Blood sample
Physical Function | 1 year
  Six-Minute Walk Test (6MWT)
Food-related aspects | 1 year
  Eating Questionnaire (EDE-Q) with 28 questions; the minimum values are 0,04 and maximum values are 4,97; Higher scores indicate greater levels of symptomatology
Anxiety and depression | 1 year
  Social appearance anxiety scale (SAAS) is a16-item self-report measure; The items on the SAAS are rated on a 5-point Likert scale, ranging from 1 (not at all) to 5 (extremely). The SAAS yields a total score, which can range from 16 to 80. Higher scores on the SAAS indicate greater social appearance anxiety.
Body image | 1 year
  Body Image Perception Questionnaire (BIQ); the 19-item Body-Image Questionnaire; The total scores range from 0 to 72 with a higher score reflecting greater impairment and likelihood
Self-Esteem | 1 year
  Coopersmith Self-Esteem Scale (CSES) The CSEI consists of 50 items and yields an overall score and four separate scores representing specific aspects of self-esteem, namely, general self, social self-peers, home parents, and school academic (or professional for adult form).
Barriers and facilitators of physical activity | 1 year
  Barriers and facilitators of physical activity Questionnaire on open questions

SECONDARY OUTCOMES:
Health-related Quality of life (IWQOL) | 1 year
  Quality of life will be assessed using the general health and well-being questionnaire; The Impact of Weight on Quality of Life-Lite (IWQOL-Lite)© is a validated, 31-item; Scores range from 0 to 100, with 100 representing the best quality of life
physical activity level | 1 year
  Activity Log App
Satisfaction with follow-up by nurses | 1 year
  Assessment Form of Nurse-led Educational Activities Satisfaction questionnaire

REFERENCES:
- [Background] Grieve E, Mackenzie RM, Munro J, O'Donnell J, Stewart S, Ali A, Bruce D, Trevor M, Logue J. Variations in bariatric surgical care pathways: a national costing study on the variability of services and impact on costs. BMC Obes. 2018 Dec 26;5:43. doi: 10.1186/s40608-018-0223-3. eCollection 2018. PMID 30607251
- [Background] Colquitt JL, Pickett K, Loveman E, Frampton GK. Surgery for weight loss in adults. Cochrane Database Syst Rev. 2014 Aug 8;2014(8):CD003641. doi: 10.1002/14651858.CD003641.pub4. PMID 25105982
- [Background] Gesquiere I, Augustijns P, Lannoo M, Matthys C, Van der Schueren B, Foulon V. Barriers in the Approach of Obese Patients Undergoing Bariatric Surgery in Flemish Hospitals. Obes Surg. 2015 Nov;25(11):2153-8. doi: 10.1007/s11695-015-1680-0. PMID 25893653
- [Background] Madsen LR, Baggesen LM, Richelsen B, Thomsen RW. Effect of Roux-en-Y gastric bypass surgery on diabetes remission and complications in individuals with type 2 diabetes: a Danish population-based matched cohort study. Diabetologia. 2019 Apr;62(4):611-620. doi: 10.1007/s00125-019-4816-2. Epub 2019 Feb 6. PMID 30734055
- [Background] Bailly L, Schiavo L, Sebastianelli L, Fabre R, Morisot A, Pradier C, Iannelli A. Preventive effect of bariatric surgery on type 2 diabetes onset in morbidly obese inpatients: a national French survey between 2008 and 2016 on 328,509 morbidly obese patients. Surg Obes Relat Dis. 2019 Mar;15(3):478-487. doi: 10.1016/j.soard.2018.12.028. Epub 2019 Jan 8. PMID 30745152
- [Background] Di Lorenzo N, Antoniou SA, Batterham RL, Busetto L, Godoroja D, Iossa A, Carrano FM, Agresta F, Alarcon I, Azran C, Bouvy N, Balague Ponz C, Buza M, Copaescu C, De Luca M, Dicker D, Di Vincenzo A, Felsenreich DM, Francis NK, Fried M, Gonzalo Prats B, Goitein D, Halford JCG, Herlesova J, Kalogridaki M, Ket H, Morales-Conde S, Piatto G, Prager G, Pruijssers S, Pucci A, Rayman S, Romano E, Sanchez-Cordero S, Vilallonga R, Silecchia G. Clinical practice guidelines of the European Association for Endoscopic Surgery (EAES) on bariatric surgery: update 2020 endorsed by IFSO-EC, EASO and ESPCOP. Surg Endosc. 2020 Jun;34(6):2332-2358. doi: 10.1007/s00464-020-07555-y. Epub 2020 Apr 23. PMID 32328827
- [Background] Mechanick JI, Apovian C, Brethauer S, Garvey WT, Joffe AM, Kim J, Kushner RF, Lindquist R, Pessah-Pollack R, Seger J, Urman RD, Adams S, Cleek JB, Correa R, Figaro MK, Flanders K, Grams J, Hurley DL, Kothari S, Seger MV, Still CD. CLINICAL PRACTICE GUIDELINES FOR THE PERIOPERATIVE NUTRITION, METABOLIC, AND NONSURGICAL SUPPORT OF PATIENTS UNDERGOING BARIATRIC PROCEDURES - 2019 UPDATE: COSPONSORED BY AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS/AMERICAN COLLEGE OF ENDOCRINOLOGY, THE OBESITY SOCIETY, AMERICAN SOCIETY FOR METABOLIC & BARIATRIC SURGERY, OBESITY MEDICINE ASSOCIATION, AND AMERICAN SOCIETY OF ANESTHESIOLOGISTS - EXECUTIVE SUMMARY. Endocr Pract. 2019 Dec;25(12):1346-1359. doi: 10.4158/GL-2019-0406. Epub 2019 Nov 4. PMID 31682518
- [Background] Petcu A. Comprehensive Care for Bariatric Surgery Patients. AACN Adv Crit Care. 2017 Fall;28(3):263-274. doi: 10.4037/aacnacc2017410. PMID 28847861
- [Background] Garcia-Delgado Y, Lopez-Madrazo-Hernandez MJ, Alvarado-Martel D, Miranda-Calderin G, Ugarte-Lopetegui A, Gonzalez-Medina RA, Hernandez-Lazaro A, Zamora G, Perez-Martin N, Sanchez-Hernandez RM, Ibarra-Gonzalez A, Bengoa-Dolon M, Mendoza-Vega CT, Appelvik-Gonzalez SM, Caballero-Diaz Y, Hernandez-Hernandez JR, Wagner AM. Prehabilitation for Bariatric Surgery: A Randomized, Controlled Trial Protocol and Pilot Study. Nutrients. 2021 Aug 24;13(9):2903. doi: 10.3390/nu13092903. PMID 34578781
- [Background] Coulman KD, Howes N, Hopkins J, Whale K, Chalmers K, Brookes S, Nicholson A, Savovic J, Ferguson Y, Owen-Smith A, Blazeby J; By-Band-Sleeve Trial Management Group; Blazeby J, Welbourn R, Byrne J, Donovan J, Reeves BC, Wordsworth S, Andrews R, Thompson JL, Mazza G, Rogers CA. A Comparison of Health Professionals' and Patients' Views of the Importance of Outcomes of Bariatric Surgery. Obes Surg. 2016 Nov;26(11):2738-2746. doi: 10.1007/s11695-016-2186-0. PMID 27138600
- [Background] Domenech-Briz V, Gomez Romero R, de Miguel-Montoya I, Juarez-Vela R, Martinez-Riera JR, Marmol-Lopez MI, Verdeguer-Gomez MV, Sanchez-Rodriguez A, Gea-Caballero V. Results of Nurse Case Management in Primary Heath Care: Bibliographic Review. Int J Environ Res Public Health. 2020 Dec 20;17(24):9541. doi: 10.3390/ijerph17249541. PMID 33419267
- [Background] Cangelosi G, Grappasonni I, Pantanetti P, Scuri S, Garda G, Cuc Thi Thu N, Petrelli F. Nurse Case Manager Lifestyle Medicine (NCMLM) in the Type Two Diabetes patient concerning post COVID-19 Pandemic management: Integrated-Scoping literature review. Ann Ig. 2022 Nov-Dec;34(6):585-602. doi: 10.7416/ai.2022.2500. Epub 2022 Feb 8. PMID 35142333
- [Result] Foreman KJ, Marquez N, Dolgert A, Fukutaki K, Fullman N, McGaughey M, Pletcher MA, Smith AE, Tang K, Yuan CW, Brown JC, Friedman J, He J, Heuton KR, Holmberg M, Patel DJ, Reidy P, Carter A, Cercy K, Chapin A, Douwes-Schultz D, Frank T, Goettsch F, Liu PY, Nandakumar V, Reitsma MB, Reuter V, Sadat N, Sorensen RJD, Srinivasan V, Updike RL, York H, Lopez AD, Lozano R, Lim SS, Mokdad AH, Vollset SE, Murray CJL. Forecasting life expectancy, years of life lost, and all-cause and cause-specific mortality for 250 causes of death: reference and alternative scenarios for 2016-40 for 195 countries and territories. Lancet. 2018 Nov 10;392(10159):2052-2090. doi: 10.1016/S0140-6736(18)31694-5. Epub 2018 Oct 16. PMID 30340847